CLINICAL TRIAL: NCT01151215
Title: A Phase II, Randomised, Double-blind, Placebo-controlled, Multi-centre Study to Assess the Efficacy and Safety of AZD8931 In Combination With Anastrozole, Compared to Anastrozole Alone, in Post Menopausal Women With Hormone Receptor Positive, Endocrine Therapy Naive, Locally Advanced or Metastatic Breast Cancer (MINT).
Brief Title: Study of Anastrozole +/- AZD8931 in Postmenopausal Women With Endocrine Therapy Naive Breast Cancer
Acronym: MINT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0102C00004
Record Dates: First submitted 2010-06-15; First posted 2010-06-28 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Neoplasms; Breast Neoplasms; Breast Cancer
Keywords: Cancer; tumour; breast cancer; metastatic; secondary; locally advanced
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Neoplasm Metastasis | interventions — AZD 8931; Anastrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): AZD8931 40mg (bd) plus anastrozole 1mg (od)
  Interventions: Drug: AZD8931; Drug: anastrozole
- 2 (Experimental): AZD8931 20mg (bd) plus anastrozole 1mg (od)
  Interventions: Drug: AZD8931; Drug: anastrozole
- 3 (Placebo Comparator): Placebo (bd) plus anastrozole 1mg (od)
  Interventions: Drug: anastrozole; Drug: Placebo

INTERVENTIONS:
Drug: AZD8931 — Tablet, oral, bd
  Arms: 1; 2
Drug: anastrozole — Tablet, oral, od
  Other Names: Arimidex
Drug: Placebo — Tablet, oral
  Arms: 3

SUMMARY:
The main purpose of this study is to compare progression free survival in patients treated with AZD8931 given in combination with anastrozole versus anastrozole alone. The secondary objective is to investigate the safety and tolerability of AZD8931 given in combination with anastrozole.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have locally advanced or metastatic breast cancer. Lesions should not be amenable to surgery or radiation of curative intent
* Hormone therapy-naive
* Estimated life expectancy of more than 12 weeks

Exclusion Criteria:

* Last dose of prior anti-cancer therapy received within 14 days (or longer if required)
* Any eye injury or corneal surgery within 3 months prior to receiving first dose of study drug.
* Currently receiving (and unwilling to discontinue) oestrogen replacement therapy. (last dose <7 days prior to randomisation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2010-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Serban Ghiorghiu, MD, Study Director — AstraZeneca; Stephen Johnston, MA, PhD, FRCP, Principal Investigator — The Royal Marsden Hospital, London
Locations (60):
- Research Site, Lake Success, New York, United States
- Brazil (6):
  - Research Site, Belo Horizonte
  - Research Site, Goiânia
  - Research Site, Ijuí
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (3):
  - Research Site, Vancouver, British Columbia
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
- Czechia (3):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Prague
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Tampere
  - Research Site, Turku
- India (6):
  - Research Site, Bangalore
  - Research Site, Hyderabad
  - Research Site, Mumbai
  - Research Site, Pune
  - Research Site, Trivandrum
  - Research Site, Vellore
- Japan (4):
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sapporo
- Mexico (4):
  - Research Site, Durango
  - Research Site, Juchitán
  - Research Site, Mérida
  - Research Site, Monterrey
- Peru (3):
  - Research Site, Callao
  - Research Site, Lima
  - Research Site, Piura
- Philippines (4):
  - Research Site, Iloilo City
  - Research Site, Lipa City
  - Research Site, Pasay
  - Research Site, Quezon City
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Elblag
  - Research Site, Krakow
  - Research Site, Warsaw
- Russia (3):
  - Research Site, Kuzmolovsky
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Africa (2):
  - Research Site, Durban
  - Research Site, Pretoria
- Research Site, Seoul, South Korea
- Research Site, Taipei, Taiwan
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Songkhla
- Ukraine (2):
  - Research Site, Dnipropetrovsk
  - Research Site, Lviv
- United Kingdom (8):
  - Research Site, Birmingham
  - Research Site, Bournemouth
  - Research Site, Coventry
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Surrey
  - Research Site, Wythenshawe, Manchester

REFERENCES:
- [Derived] Johnston S, Basik M, Hegg R, Lausoontornsiri W, Grzeda L, Clemons M, Dreosti L, Mann H, Stuart M, Cristofanilli M. Inhibition of EGFR, HER2, and HER3 signaling with AZD8931 in combination with anastrozole as an anticancer approach: Phase II randomized study in women with endocrine-therapy-naive advanced breast cancer. Breast Cancer Res Treat. 2016 Nov;160(1):91-99. doi: 10.1007/s10549-016-3979-5. Epub 2016 Sep 21. PMID 27654971

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 482 patients were enrolled into the study, of these, 123 patients failed screening and 359 patients were randomized, 120 to AZD8931 40mg(bd) plus anastrozole 1mg (od), 118 to AZD8931 20mg(bd) plus anastrozole 1mg (od) and 121 to placebo(bd) plus anastrozole 1mg(od)
Groups:
- AZD8931 40mg + Anastrozole 1mg: AZD8931 40mg (bd) plus anastrozole 1mg (od)
- AZD8931 20mg + Anastrozole 1mg: AZD8931 20mg (bd) plus anastrozole 1mg (od)
- Placebo + Anastrozole 1mg: Placebo (bd) plus anastrozole 1mg (od)
Period: Overall Study
Arm/Group | AZD8931 40mg + Anastrozole 1mg | AZD8931 20mg + Anastrozole 1mg | Placebo + Anastrozole 1mg
Started | 120 | 118 | 121
Completed | 100 (This is number of patients who were continuing at cut off (ie not withdrawn)) | 95 (This is number of patients who were continuing at cut off (ie not withdrawn)) | 102 (This is number of patients who were continuing at cut off (ie not withdrawn))
Not Completed | 20 | 23 | 19
Not completed — Worsening of condition under study | 1 | 1 | 1
Not completed — Death | 16 | 20 | 11
Not completed — Lost to Follow-up | 0 | 0 | 3
Not completed — Withdrawal by Subject | 3 | 1 | 2
Not completed — Disease progression | 0 | 1 | 1
Not completed — Safety as judged by the investigator | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD8931 40mg + Anastrozole 1mg | AZD8931 20mg + Anastrozole 1mg | Placebo + Anastrozole 1mg | Total
Number analyzed (Participants) | 120 | 118 | 121 | 359
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (10.69) | 62.0 (11.23) | 60.5 (10.29) | 61.0 (10.73)
Sex/Gender, Customized [Number; unit: Participants] — Female only
  Participants | 120 | 118 | 121 | 359
Race/Ethnicity, Customized [Number; unit: Participants]
  Ethnicity: Hispanic or Latino | 51 | 53 | 45 | 149
  Ethnicity: Native American | 1 | 0 | 0 | 1
  Ethnicity: African | 2 | 1 | 4 | 7
  Ethnicity: Asian (other than Chinese/Japanese) | 35 | 31 | 32 | 98
  Ethnicity: Chinese | 0 | 0 | 1 | 1
  Ethnicity: Japanese | 0 | 5 | 3 | 8
  Ethnicity: Other | 12 | 17 | 17 | 46
  Ethnicity: Not applicable | 19 | 11 | 19 | 49
Race/Ethnicity, Customized [Number; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Asian | 35 | 37 | 36 | 108
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Black or African American | 5 | 7 | 6 | 18
  Race: White | 50 | 56 | 60 | 166
  Race: Other | 30 | 18 | 19 | 67
Study Stratification: Disease Classification [Number; unit: Participants] — Study was stratified by locally advanced / metastatic disease
  Participants
    Locally advanced | 28 | 27 | 28 | 83
    Metastatic disease | 92 | 91 | 93 | 276

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival as Evaluated by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
Description: Time from the date of randomization until the date of objective disease progression (as per RECIST 1.1) or the date of death (by any cause in the absence of progression). Disease progression is defined using RECIST 1.1 as >=20% increase in the sum of longest diameters of target lesions and an absolute increase of >=5mm, taking as reference the smallest sum of longest diameters of target lesions since study start, or unequivocal progression in non-target lesions, or appearance of any new lesions.
Time Frame: Tumour assessment by RECIST 1.1 every 12 weeks until data cut-off at 31 August 2012
Population: Full Analysis Set (all participants randomized, irrespective of whether treatment was received). Participants are analysed according to the treatment group they were randomized to.
Measure: Median (Inter-Quartile Range); unit: Months
Units Other Than Participants: Events
Arm/Group | AZD8931 40mg + Anastrozole 1mg | AZD8931 20mg + Anastrozole 1mg | Placebo + Anastrozole 1mg
Number analyzed (Participants) | 120 | 118 | 121
Number analyzed (Events) | 47 | 49 | 45
Months | 13.8 [5.5 to 22.1] | 10.9 [5.4 to NA] — Upper limit of inter-quartile range is not calculable | 14.0 [6.7 to 21.8]
Statistical Analysis 1: Comparison: AZD8931 40mg + Anastrozole 1mg vs Placebo + Anastrozole 1mg; 345 patients were to be randomised to observe at least 233 progression events, based on HR=0.60, 90% power, 2-sided 5% significant level and a median of 9 months for the placebo arm. An interim analysis with futility boundary was introduced based on an IDMC recommendation; Test type: Superiority or Other; p = 0.485, Log Rank — Statistical significance threshold at this interim analysis was 5%; The log rank test was stratified for the IVRS stratification factor of disease classification (locally advanced / metastatic disease); Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.77 to 1.75] — The Hazard Ratio is for AZD8931 40mg + anastrozole 1mg / Placebo + anastrozole 1mg, ie a hazard ratio <1 favours AZD8931 40mg + anastrozole 1mg
Statistical Analysis 2: Comparison: AZD8931 20mg + Anastrozole 1mg vs Placebo + Anastrozole 1mg; 345 patients were to be randomised to observe at least 233 progression events, based on HR=0.6, 90% power, 2-sided 5% significant level and a median of 9 months for the placebo arm. An interim analysis with futility boundary was introduced based on an IDMC recommendation; Test type: Superiority or Other; p = 0.135, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.37, 95% CI 2-sided [0.91 to 2.06] — The Hazard ratio is for AZD8931 20mg + anastrozole 1mg / Placebo + anastrozole 1mg, ie a hazard ratio < 1 favours AZD8931 20mg + anastrozole 1mg

2. Secondary Outcome: Compare the Overall Survival in Patients Treated With AZD8931 in Combination With Anastrozole Versus Anastrozole Alone
Description: Time from the date of randomization to the date of death (by any cause)
Time Frame: Following progression, patients were contacted at 12 weekly intervals until data cut-off at 31 August 2012 to determine survival status
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Months
Units Other Than Participants: Events
Arm/Group | AZD8931 40mg + Anastrozole 1mg | AZD8931 20mg + Anastrozole 1mg | Placebo + Anastrozole 1mg
Number analyzed (Participants) | 120 | 118 | 121
Number analyzed (Events) | 16 | 20 | 12
Months | 6.9 [4.6 to 14.3] | 8.3 [4.7 to 14.0] | 7.9 [4.6 to 14.5]

ADVERSE EVENTS:
Arm/Group | AZD8931 20mg | AZD8931 40mg | Placebo
Serious Adverse Events (participants affected / at risk) | 14/118 | 17/120 | 11/121
Other Adverse Events (participants affected / at risk) | 112/118 | 115/120 | 99/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8931 20mg (N=118) | AZD8931 40mg (N=120) | Placebo (N=121)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
COR PULMONALE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
CEREBELLAR INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
COMA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MONOPARESIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
BREAST HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8931 20mg (N=118) | AZD8931 40mg (N=120) | Placebo (N=121)
ANAEMIA (Blood and lymphatic system disorders) | 7 (7) | 10 (10) | 6 (6)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 1 (1)
CHEST PAIN (General disorders) | 3 (3) | 1 (1) | 0 (0)
MUCOSAL DRYNESS (General disorders) | 1 (1) | 2 (2) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 10 (10) | 5 (6) | 7 (7)
PAIN (General disorders) | 2 (2) | 3 (3) | 2 (2)
PYREXIA (General disorders) | 3 (4) | 8 (9) | 5 (11)
SPINAL PAIN (General disorders) | 2 (2) | 0 (0) | 1 (1)
SWELLING (General disorders) | 2 (2) | 0 (0) | 1 (1)
XEROSIS (General disorders) | 0 (0) | 4 (4) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
PARONYCHIA (Infections and infestations) | 6 (9) | 22 (26) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 2 (2) | 1 (1) | 0 (0)
WEIGHT INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 8 (9)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 4 (4)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 4 (8) | 11 (11) | 4 (4)
DEPRESSION (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
BLISTER (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 3 (3)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
BLEPHARITIS (Eye disorders) | 2 (2) | 4 (7) | 0 (0)
DRY EYE (Eye disorders) | 5 (5) | 8 (8) | 2 (2)
EYE PAIN (Eye disorders) | 2 (2) | 0 (0) | 2 (3)
VITREOUS FLOATERS (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 4 (5) | 11 (11) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
ASTHENIA (General disorders) | 4 (5) | 7 (8) | 9 (9)
OEDEMA (General disorders) | 1 (1) | 4 (4) | 0 (0)
BREAST INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
FUNGAL INFECTION (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 3 (3) | 4 (4) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 14 (15) | 10 (10) | 12 (13)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
INSOMNIA (Psychiatric disorders) | 4 (4) | 4 (5) | 11 (12)
DYSURIA (Renal and urinary disorders) | 3 (3) | 5 (11) | 0 (0)
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (12) | 6 (6)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 5 (6)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 6 (6) | 9 (9) | 5 (5)
DRY SKIN (Skin and subcutaneous tissue disorders) | 22 (24) | 30 (32) | 3 (3)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
NAIL RIDGING (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
PAPULE (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
LYMPHOEDEMA (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
PALPITATIONS (Cardiac disorders) | 0 (0) | 4 (4) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2)
CONJUNCTIVITIS (Eye disorders) | 6 (7) | 10 (13) | 2 (2)
EYE IRRITATION (Eye disorders) | 2 (2) | 7 (9) | 1 (1)
EYE PRURITUS (Eye disorders) | 6 (7) | 3 (3) | 4 (4)
OCULAR HYPERAEMIA (Eye disorders) | 1 (1) | 2 (2) | 2 (2)
VISION BLURRED (Eye disorders) | 1 (1) | 4 (4) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (5) | 8 (10) | 9 (9)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 (5) | 6 (6) | 8 (8)
CONSTIPATION (Gastrointestinal disorders) | 6 (6) | 5 (5) | 7 (8)
DIARRHOEA (Gastrointestinal disorders) | 46 (70) | 61 (103) | 13 (16)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 13 (18) | 16 (20) | 12 (14)
STOMATITIS (Gastrointestinal disorders) | 6 (6) | 9 (9) | 4 (4)
TONGUE ULCERATION (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 9 (10) | 13 (16) | 11 (12)
FATIGUE (General disorders) | 11 (11) | 8 (9) | 11 (11)
FEELING COLD (General disorders) | 2 (2) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 2 (2)
IRRITABILITY (General disorders) | 0 (0) | 0 (0) | 2 (2)
MUCOSAL INFLAMMATION (General disorders) | 6 (8) | 10 (13) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2) | 2 (2) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
CELLULITIS (Infections and infestations) | 3 (4) | 2 (2) | 1 (1)
CYSTITIS (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
FOLLICULITIS (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
FURUNCLE (Infections and infestations) | 0 (0) | 2 (4) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
NAIL INFECTION (Infections and infestations) | 2 (2) | 1 (3) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 3 (4) | 7 (8) | 2 (2)
ONYCHOMYCOSIS (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
RASH PUSTULAR (Infections and infestations) | 7 (9) | 15 (17) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (2) | 3 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (5) | 3 (3) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 11 (13) | 13 (15) | 10 (15)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3) | 5 (7) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (5) | 6 (6) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 3 (3) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 3 (4) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 2 (2) | 9 (10) | 4 (5)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3 (3) | 5 (5) | 2 (2)
DECREASED APPETITE (Metabolism and nutrition disorders) | 14 (16) | 11 (11) | 5 (5)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 14 (15) | 10 (10) | 23 (27)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7) | 6 (6)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 6 (7) | 5 (5) | 5 (5)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 9 (9)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 13 (15) | 5 (5) | 7 (10)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (2) | 0 (0)
AGEUSIA (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 10 (12) | 10 (13) | 18 (23)
LETHARGY (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
ANXIETY (Psychiatric disorders) | 2 (2) | 1 (1) | 4 (5)
MOOD SWINGS (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
LEUKOCYTURIA (Renal and urinary disorders) | 1 (2) | 5 (6) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 4 (4) | 6 (6) | 6 (15)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 2 (2)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6) | 0 (0)
NASAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
ACNE (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (9) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6) | 0 (0)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 19 (23) | 31 (37) | 2 (2)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (9) | 3 (15)
NAIL DYSTROPHY (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 3 (3) | 13 (13) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 15 (17) | 10 (13) | 4 (4)
RASH (Skin and subcutaneous tissue disorders) | 38 (42) | 56 (78) | 15 (20)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (7) | 2 (2)
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 1 (1)
HOT FLUSH (Vascular disorders) | 4 (4) | 1 (1) | 11 (11)
HYPERTENSION (Vascular disorders) | 7 (8) | 9 (10) | 3 (6)

LIMITATIONS AND CAVEATS:
The final analysis for this study is the analysis that was sent to the study's IDMC, based on a data cut-off of 31 August 2012. At the data cut-off point the data was cleaned, but 9 adverse events were not coded. These events are not included here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days